CLINICAL TRIAL: NCT05510427
Title: Phase Ib Trial of Infigratinib In Combination With Atezolizumab And Bevacizumab for The Second-Line Treatment of Advanced Cholangiocarcinoma With FGFR2 Fusion/Amplification
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Per PI's request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0149; NCI-2022-06868 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Cholangiocarcinoma; Liver Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Liver Neoplasms | interventions — infigratinib; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Dose Escalation) (Experimental): The first group of participants will receive the lowest dose level of infigratinib.
  Interventions: Drug: Infigratinib; Drug: Atezolizumab; Drug: Bevacizumab
- Part B (Dose Expansion) (Experimental): Participants will receive infigratinib at the recommended dose that was found in Part A.
  Interventions: Drug: Infigratinib; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Infigratinib — Given by PO
Drug: Atezolizumab — Given by (IV) vein
Drug: Bevacizumab — Given by (IV) vein

SUMMARY:
To find the highest tolerable dose of infigratinib that can be given in combination with bevacizumab and atezolizumab to patients with advanced/metastatic CCA with a FGFR2 mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE(S):

• To determine the safety and maximum tolerated dose (MTD) of the triple combination of infigratinib with bevacizumab and atezolizumab in patients with FGFR-altered metastatic CCA.

SECONDARY OBJECTIVE(S):

* To determine the overall response rate (ORR), as assessed by the treating Investigator according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* To evaluate the duration of response in subjects with best overall response of complete response (CR) or partial response (PR).
* To evaluate PFS defined as the time from the start of study treatment to disease progression or death, whichever occurs first.
* To evaluate the duration of OS defined as the time from the start of study treatment to death from any cause.
* To evaluate the clinical benefit rate defined as the proportion of subjects with best overall response of CR, PR, or stable disease

EXPLORATORY OBJECTIVE:

• To examine the change of the immune microenvironment with this treatment combination in tumor and blood samplesusing a validated immune biomarker panel and liquid biopsy (end-of-treatment genomic markers using cfDNA analysis) to study resistance to infigratinib and identify response markers from trial medications.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged ≥18 years.
2. Has histologically confirmed metastatic or advanced unresectable cholangiocarcinoma.
3. Has disease that is measurable per the RECIST v1.1.
4. Has FGFR2 fusion in tumor tissue. Presence of the FGFR2 fusion should be determined by CLIA-validated genomic testing of a tumor tissue specimen (DNA-based or RNA-based).
5. Is refractory to, has demonstrated intolerance to, or has refused access to, available standard therapies. Refractory patients should have evidence of progressive disease on at least one prior standard chemotherapy regimen for advanced or metastatic disease. Patients who discontinued available standard therapy due to toxicity must have continued evidence of measurable disease.
6. Has archival formalin-fixed, paraffin-embedded primary tumor tissue available or patient is willing to undergo a pretreatment biopsy.
7. Is able to take oral medication.
8. Is able to comply with protocol procedures and scheduled visits.
9. Has Eastern Cooperative Oncology Group performance status of 0 or 1
10. Has adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

    * Absolute neutrophil count (ANC) ≥ 1.0 × 109/L (1000/µL) without granulocyte colony-stimulating factor support
    * Platelet count ≥ 75 × 109/L (75,000/µL) without transfusion
    * Hemoglobin ≥ 80 g/L (8 g/dL) i. Patients may be transfused to meet this criterion.
    * Aspartate amino transferate (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × upper limit of normal (ULN), with the following exceptions: i. Patients with documented liver metastases: AST and ALT

      * 5 × ULN ii. Patients with documented liver or bone metastases: ALP
      * 5 × ULN
    * Serum bilirubin ≤ 1.5 × ULN with the following exception:

      i. Patients with known Gilbert disease: serum bilirubin

      ≤ 3 × ULN
    * Serum creatinine ≤ 1.5 × ULN
    * Serum albumin ≥ 25 g/L (2.5 g/dL)
    * For patients not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
11. Has a negative human immunodeficiency virus (HIV) test at screening with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200 and have an undetectable viral load
12. Has a negative hepatitis B surface antigen (HBsAg) test at screening (unless patient has chronic HBV on anti viral therapy)
13. Has a negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening (unless patient has chronic HBV on anti viral therapy) The HBV DNA test will be performed only for patients who have a negative HBsAg test and a positive total HBcAb test. Patients with chronic HBV on antiviral therapy or HCV patients who have completed curative anti-viral therapy can be included.
14. The effects of the proposed bevacizumab+atezolizumab+infigratinib combination on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation (refer to MDA Policy CLN 1114), and for 6 months after the last study drug dose. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months)
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy)
    * History of bilateral tubal ligation or another surgical sterilization procedure. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
15. Men treated or enrolled on this protocol must also agree to use adequate contraception and agree to to refrain from donating sperm prior to the study, for the duration of study participation, and 6 months after completion of bevacizumab+atezolizumab+infigratinib administration.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Patients with untreated CNS metastases are excluded from study

   * Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
   * Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:
   * Measurable disease, per RECIST v1.1, must be present outside the CNS.
   * The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
   * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
   * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease.
   * If the patient is receiving anti-convulsant therapy, the dose is considered stable. IF BRAIN SCANS are not done: Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
   * There is no evidence of interim progression between completion of CNS directed therapy and initiation of study treatment.
   * Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy and/or surgery, with no need to repeat the screening brain scan.
2. Received treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, or anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipates a need for systemic immunosuppressive medication during study treatment, with the following exceptions:

   * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
3. Received chemotherapy, biologic therapy, immunotherapy, or investigational agent within 4 weeks prior to enrollment.
4. Received treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
5. Had previous treatment with any of the following:

   * selective FGFR inhibitors or immune-checkpoint inhibitors.
   * any VEGFR-targeting agent targeting including bevacizumab, ramucirumab, pazopanib, and other anti-angiogenesis inhibitors.
   * CD137 agonists or immune checkpoint-blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
6. Has a history and/or has current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, vascular system, and lung. Exceptions include calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcifications-these are allowed.
7. Has history or current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, inflammation or ulceration, keratoconjunctivitis, or diabetic retinopathy, confirmed by ophthalmic physician. Subjects with asymptomatic ophthalmic conditions assessed by the investigator to pose minimal risk for study participation may be enrolled in the study.
8. Are currently receiving or are planning to receive during participation in this study, treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs, including carbamazepine, phenytoin, phenobarbital, and primidone.
9. Have consumed grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges or products containing juice of these fruits within 7 days prior to first dose of study drug.
10. Had a gastrointestinal bleed requiring transfusion or invasive intervention within 3 months prior to enrollment.
11. Has a history of deep vein thrombosis, pulmonary embolism, or any other thromboembolism, including portal venous thrombosis within 3 months prior to enrollment. Venous port or catheter thrombosis, incidental asymptomatic pulmonary embolism diagnosed on imaging studies, or superficial venous thrombosis are not considered significant and are allowed. Has current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants (including direct oral anticoagulants); thrombolytic agents for therapeutic (as opposed to prophylactic) purpose; use of aspirin (> 325 mg/day); or use of clopidogrel (> 75 mg/day). Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR <1.5 ULN and an activated partial thromboplastin time (aPTT) within normal limits within 14 days prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa) and rivaroxaban (Xarelto) is not recommended due to bleeding risk.
12. Had a history of any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina within 6 months prior to enrollment.
13. Has a history of uncontrolled or poorly-controlled hypertension (>150 mmHg systolic or >100 mmHg diastolic), hypertensive crisis or hypertensive encephalopathy
14. Had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment.
15. Had a major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipates need for a major surgical procedure during the study

    • Note: Placement of a vascular access device should be at least 2 days prior to initiation of study treatment
16. Is receiving chronic antiplatelet therapy, nonsteroidal anti-inflammatory drugs (e.g., ibuprofen, naproxen), dipyridamole, clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is allowed.
17. Has had significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization
18. Has a history of central nervous system disease or evidence of this disease upon physical or neurological examination.
19. Has a history of moderate to severe hemoptysis (defined as ≥ 2.5 mL of bright red blood per episode) within 1 month prior to screening
20. Has a history or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
21. Has a history of abdominal fistula, gastrointestinal (GI) perforation, intraabdominal abscess, or active GI bleeding within 6 months prior to randomization
22. Serious, non-healing wound, active ulcer, or untreated bone fracture
23. Had a history of malignancy other than cholangiocarcinoma within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
24. Has a history of leptomeningeal disease
25. Has uncontrolled tumor-related pain

    * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should have recovered from the effects of radiation. There is no required minimum recovery period.
    * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy, if appropriate, prior to enrollment.
26. Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (at a frequency of at least once monthly)

    * Patients with indwelling catheters (e.g., PleurX) are allowed.
27. Has uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL, or corrected serum calcium > ULN)

29. Has current evidence of endocrine alterations of calcium/phosphate homeostasis, eg, parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis, and other disorders. 30. Has elevated phosphorus or abnormal serum calcium, or phosphorus, or calcium-phosphorus product ≥ 55 mg2/dL2:

a. Inorganic phosphorus > 1.02 × ULN b. Total corrected serum calcium > 1.02 × ULN or < 1.02 × LLN 31.Has active or a history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

* Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
* Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met: i. Rash must cover < 10% of body surface area ii. Disease is well controlled at baseline and requires only lowpotency topical corticosteroids iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet-A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months 32.Has a history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis; or has evidence of active pneumonitis upon screening via computed tomography (CT) scan of the chest

  a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted. 33.Had significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident); unstable arrhythmia; or unstable angina within 3 months prior to initiation of study treatment 34.Had a severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, including COVID-19, bacteremia, active tuberculosis or severe pneumonia. 35.Received treatment with therapeutic oral- or IV antibiotics within 2 weeks prior to initiation of study treatment
* Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study. 36.Had a prior allogeneic stem cell or solid organ transplantation 37.Has any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that may render the patient at high risk from treatment complications 38.Received treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipates need for such a vaccine during treatment or within 5 months after the final dose of treatment. Receipt of SARS-CoV vaccine is allowed. 39.Has a history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins 40.Has a known allergy or hypersensitivity to any component of the infigratinib, bevacizumab, or atezolizumab formulations 41.Is pregnant or breastfeeding, or intention of becoming pregnant during study treatment or within 6 months after the final dose of study treatment Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Sunyoung Lee, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org